CLINICAL TRIAL: NCT01103180
Title: SSRIs and Self-harm in Borderline Personality Disorder
Brief Title: Selective Serotonin Reuptake Inhibitors (SSRIs) in Borderline Personality Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn due to inability to accrue
Sponsor: University of Chicago (Other)
Collaborators: Temple University (Other); Northwestern University (Other); University of Southern Mississippi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH084904
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Borderline Personality Disorder
Keywords: Selective Serotonin Reuptake Inhibitor; Escitalopram; Borderline Personality Disorder; Major Depressive Disorder; Self-harm
MeSH Terms: conditions — Borderline Personality Disorder; Depressive Disorder, Major; Self-Injurious Behavior | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): 10-20 mg of escitalopram for eight weeks (10mg for the first 2 weeks, 20mg thereafter)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Inert placebo (sugar pill) taken daily for eight weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10-20 mg of escitalopram daily for eight weeks (10mg for the first 2 weeks, 20mg thereafter)
  Other Names: Lexapro

SUMMARY:
The goal of this study is to examine the effectiveness the selective serotonin reuptake inhibitor (SSRI) escitalopram (also known by the trade name "Lexapro") in reducing desire to self-harm and actual self-harming among young adults with borderline personality disorder who are also currently depressed. Subjects will receive either escitalopram or placebo for eight weeks. During this time subjects will be make weekly visits to see the psychiatrist and record their thoughts and feelings several times each day using an electronic diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Borderline Personality Disorder
* Current Major Depression

Exclusion Criteria:

* Past 2 months SSRI use
* Past 6 months non-SSRI antidepressant use
* Past 2 months initiation of psychotherapy
* Lifetime bipolar disorder, organic disorder, psychotic disorder
* Current alcohol or drug dependence
* Current severe suicidal / homicidal ideation necessitating immediate medical intervention
* Currently pregnancy or nursing
* Unable or unwilling to cooperate with study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S McCloskey, Ph.D, Principal Investigator — Temple University (primary) / University of Chicago; Emil F Coccaro, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Hospitals, Chicago, Illinois, United States

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 35 | 35
Completed | 13 | 14
Not Completed | 22 | 21
Not completed — Withdrawal by Subject | 8 | 13
Not completed — Lost to Follow-up | 13 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (9.9) | 27.3 (8.8) | 28.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Self-harm Ideation
Description: Self-harm ideation was measured by electronic diaries (EMA) up to four times a day. Each time a person completed an EMA diary they were asked to rate their urge to hurt themselves on a 5 point scale ( 0 to 4) pad where 0 is not at all, 2 is moderately and 4 is extremely strong.
Time Frame: pre-treatment (week 0) to post-treatment (end of week 8)
Population: Data was not collected because the study was terminated.
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms was assessed via (a) electronic diary (i.e. sum of eight POMS-D items: sad, unhappy, blue, hopeless, discouraged, miserable, helpless and worthless rated using 0-4 scale above) and (b) weekly interview(Hamilton depression rating)
Time Frame: baseline (week 0) and post treatment (week 8).
Population: Data was not collected because the study was terminated.
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
Early study termination due to recruitment difficulties leading to none of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No